CLINICAL TRIAL: NCT03433807
Title: Expanded Access Protocol (EAP) of Idebenone in Patients With Duchenne Muscular Dystrophy
Brief Title: Expanded Access Program for Idebenone in Participants With Duchenne Muscular Dystrophy (DMD)
Status: No longer available | Type: Expanded Access
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SNT-EAP-002
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: idebenone, DMD, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — idebenone

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Idebenone — 900 mg idebenone/day (2 tablets to be taken 3 times a day with meals)

SUMMARY:
The primary objective of this Expanded Access Program is to provide idebenone as a treatment for eligible participants with Duchenne Muscular Dystrophy before it is commercially available in the United States (U.S.) for the indication of DMD.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of DMD (severe dystrophinopathy) and clinical features consistent of typical DMD at diagnosis (i.e., documented delayed motor skills and muscle weakness by age 5 years) and who in the opinion of the Treating physician would benefit from treatment with idebenone. DMD should be confirmed by mutation analysis in the dystrophin gene or by substantially reduced levels of dystrophin protein (i.e., absent or <5% of normal) on Western blot or immunostaining.
* Minimum 8 years old at Prescreening.
* PEF or FVC ≤80% and >25% of predicted value based on most recent assessment noted in the patient's medical record and subsequently confirmed at the Enrollment Visit.
* Able to understand program requirements and swallow program medication.
* Signed and dated Informed Consent Form (to be obtained at the Enrollment Visit from patient or parent/legal guardian (if applicable) prior to performing any program-specific procedures and dispensing idebenone to the patient).

Exclusion Criteria:

* Eligible for and able to participate in an ongoing clinical trial of idebenone.
* Is at high-risk of a fatal outcome from lung infection and/or advanced cardiomyopathy in the opinion of the Treating physician.
* Known moderate or severe impairment of hepatic function or severe impairment of renal function.
* Prior or ongoing medical condition or laboratory abnormality which in the Treating physician's opinion may put the patient at significant risk or may interfere significantly with the patient's participation in the program.
* Abuse of drugs or alcohol, which in Treating physician's opinion would interfere with the compliance to treatment.
* Known individual hypersensitivity to idebenone or to any of the ingredients/excipients of the program medication.

Min Age: 8 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger, Baltimore, Maryland
  - Columbia University Pediatric Neuromuscular Center, New York, New York
  - Carolina's Healthcare System, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - St. Luke's Rehabilitation Institute, Spokane, Washington